CLINICAL TRIAL: NCT01203891
Title: Single Photon Emission Computed Tomography of the Normal Human Brain
Status: Completed | Type: Observational
Sponsor: Amen Clinics, Inc. (Industry)
Responsible Party: Dr. Daniel Amen, Amen Clinics, Inc.
Other Study IDs: 20021714
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Normal Human Subjects
Keywords: SPECT; Imaging; Healthy brain; regional cerebral blood flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy brain subjects: The study seeks to recruit 100 normal, healthy brain subjects between ages 10 and 90 for SPECT brain imaging.

SUMMARY:
The objective of the study is to acquire a database of Single Photon Emission Computed Tomographic (SPECT) studies of the brains of normal human subjects in resting and concentrating states. The database will provide a basis for subsequent investigation of meaningful brain differences between clinical and normal subject groups

DETAILED DESCRIPTION:
See brief summary.

ELIGIBILITY:
Inclusion Criteria:

The study seeks to recruit 100 normal human subjects between ages 10 and 90 for SPECT brain imaging. Subjects will initially be screened for psychiatric and other major illnesses with a screening questionnaire; they will also be given a standard DSM-4 computer-administered questionnaire (The DISC for children and teens and the SCID for adults). They will also meet individually with a psychiatrist or psychological assistant for a screening interview.

Exclusion Criteria:

1. Suicidal thinking or behavior
2. Any psychiatric diagnosis assignable under contemporary DSM nosology
3. Unstable medical condition
4. epilepsy, serious head injury, or other significant neurological disorder or use of central nervous system medication.
5. Dementia, mental retardation, or coma
6. Substance abuse or alcoholism
7. Unreliability or inability to adhere to the requirements of the study
8. Inability to personally tolerate the requirements of the study
9. Significant exposure to occupational, diagnostic, or therapeutic radiation within the prior year
10. Pregnancy or breast-feeding
11. A first-degree relative meeting any of criteria 1 through 6.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study seeks to recruit 100 subjects between ages 10 and 90 for SPECT brain imaging.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2003-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Baseline SPECT image | 24 hour assessment and data may be presented up to 10 years later as part of a normative database
  For the baseline resting study with adult subjects approximately 20 milliCuries of Tc-99m-hexamethylpropylene amine oxime (HMPAO, commercially marketed by Amersham Pharmaceuticals under the trade name Ceretec) will be injected after the initial equilibration period. Ceretec is an FDA-approved functional brain imaging radiopharmaceutical currently widely commercially available.

SECONDARY OUTCOMES:
Concentration SPECT image | 24 hour assessment and data may be presented up to 10 years later as part of a normative database
  For the concentration study the subject will start the Conner's Continuous Performance Task, a 15-minute computer-administered test of attention, subsequent to the accommodation period. Three minutes into task performance HMPAO will be injected through the catheter with attention to minimal disruption of the subject's attention task. The subject will proceed to completion of the attention task.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Amen, MD, Principal Investigator — Amen Clinics, Inc.
Locations (1):
- Amen Clinics, Inc., Newport Beach, California, United States